CLINICAL TRIAL: NCT02297763
Title: Prophylactic Quetiapine on Delirium Prevention in Critically Ill Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: YJLSM2014
Record Dates: First submitted 2014-07-04; First posted 2014-11-21 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-07

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- quetiapine (Active Comparator): quetiapine 12.5mg (bwt <50kg ) or 25mg (bwt>= 50kg) study medicine is pulverized to power and melted in 10cc tepid water. The study medicine(quetiapine) will be provided as liquid form.
  Interventions: Drug: quetiapine
- placebo (Placebo Comparator): The placebo is made of 100mg of corn starch which is melted in 10cc water.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: quetiapine — patient body weight <50kg : quetiapine 12.5mg patient body weight >=50kg : quetiapine 25mg
  quetiapine 12.5mg (bwt <50kg ) or 25mg (bwt>= 50kg) study medicine is pulverized to power and melted in 10cc tepid water. The study medicine(quetiapine) will be provided as liquid form.
  The study medicine(quetiapine) was provided as liquid form (medicine was pulverized and melted in 10cc water).
  Arms: quetiapine
Drug: placebo — The placebo is made of 100mg of corn starch which is melted in 10cc water.
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of low dose quetiapine for the prophylaxis of delirium in critically ill patients in medical intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 19 years of age, admitting to medical ICU, anticipated to stay more than 72hours

Exclusion Criteria:

* Female patients who are pregnant or breastfeeding
* active delirium
* Received other anti-psychotic drug before attend the study
* severe bradycardia
* alcohol intoxication
* No written consent from the legal representatives
* Being ill with renal or hepatic failure

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Development of delirium within 14 days after admitting to ICU (Rate) | 14 days after admitting to intensive care unit

SECONDARY OUTCOMES:
Duration of delirium occurring within 14 days after admitting to ICU (Days) | 14 days after admitting to ICU
Length of stay in ICU and hospital (Days) | up to 24 weeks
60 days in hospital mortality (Rate) | 60 days after admitting to ICU
Duration of mechanical ventilation in ICU (Days) | 14days after admitting to intensive care unit